CLINICAL TRIAL: NCT03737318
Title: Correcting Residual Errors With Spectral, Ultrasound, and Traditional Speech Therapy: A Randomized Controlled Trial
Brief Title: Correcting Residual Errors With Spectral, Ultrasound, Traditional Speech Therapy
Acronym: C-RESULTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Syracuse University (Other); Montclair State University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-RESULTS-RCT; R01DC017476 (NIH)
Record Dates: First submitted 2018-10-31; First posted 2018-11-09 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-03

CONDITIONS: Speech Sound Disorder
Keywords: speech, articulation, motor development
MeSH Terms: conditions — Speech Sound Disorder; Speech

STUDY DESIGN:
Intervention Model Description: All participants will complete a Dynamic Assessment session (Phase 0) consisting of 2 hours of traditional (non-biofeedback) instruction. Participants will be categorized into high, moderate, and low response groups based on performance in Phase 0, and the response groups will be block randomized to traditional or biofeedback speech treatment. Within the biofeedback condition, individuals will be sub-randomized in equal numbers to receive visual-acoustic or ultrasound treatment. Participants will then complete two phases of speech treatment in their randomly assigned condition. Phase 1 (Acquisition) will consist of high-intensity, highly interactive practice delivered in three 90-minute sessions over one week. Phase 2 (Generalization) will elicit structured practice of /r/ in 16 semiweekly 45-minute sessions over 8 weeks.
Who Masked: Outcomes Assessor
Masking Description: All perceptual ratings will be obtained from blinded, naive listeners recruited through online crowdsourcing. Following protocols refined in previous published research, binary rating responses will be aggregated over at least 9 unique listeners per token.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Traditional articulation treatment
  Interventions: Behavioral: Traditional articulation treatment
- Group 2 (Experimental): Biofeedback--visual-acoustic
  Interventions: Behavioral: Biofeedback--visual-acoustic; Behavioral: Traditional articulation treatment
- Group 3 (Experimental): Biofeedback-ultrasound
  Interventions: Behavioral: Biofeedback-ultrasound; Behavioral: Traditional articulation treatment

INTERVENTIONS:
Behavioral: Biofeedback-ultrasound — In ultrasound biofeedback, the elements of traditional treatment (auditory models and verbal descriptions of articulator placement) are enhanced with a real-time ultrasound display of the shape and movements of the tongue. One or two target tongue shapes will be selected for each participant, and a trace of the selected target will be superimposed over the ultrasound screen. Participants will be cued to reshape the tongue to match this target during /r/ production.
  Arms: Group 3
Behavioral: Biofeedback--visual-acoustic — In visual-acoustic biofeedback treatment, the elements of traditional treatment (auditory models and verbal descriptions of articulator placement) are enhanced with a dynamic display of the speech signal in the form of the real-time LPC (Linear Predictive Coding) spectrum. Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. They will be encouraged to attend to the visual display while adjusting the placement of their articulators and observing how those adjustments impact F3.
  Arms: Group 2
Behavioral: Traditional articulation treatment — Traditional articulation treatment involves providing auditory models and verbal descriptions of correct articulator placement, then cueing repetitive motor practice. Images and diagrams of the vocal tract will be used as visual aids; however, no real-time visual display of articulatory or acoustic information will be made available.

SUMMARY:
Children with speech sound disorder show diminished accuracy and intelligibility in spoken communication and may thus be perceived as less capable or intelligent than peers, with negative consequences for both socioemotional and socioeconomic outcomes. While most speech errors resolve by the late school-age years, between 2-5% of speakers exhibit residual speech errors (RSE) that persist through adolescence or even adulthood, reflecting about 6 million cases in the US. Both affected children/families and speech-language pathologists (SLPs) have highlighted the critical need for research to identify more effective forms of treatment for children with RSE. In a series of single-case experimental studies, research has found that treatment incorporating technologically enhanced sensory feedback (visual-acoustic biofeedback, ultrasound biofeedback) can improve speech in individuals with RSE who have not responded to previous intervention. A randomized controlled trial (RCT) comparing traditional vs biofeedback-enhanced intervention is the essential next step to inform evidence-based decision-making for this prevalent population. Larger-scale research is also needed to understand heterogeneity across individuals in the magnitude of response to biofeedback treatment.

The overall objective of this proposal is to conduct clinical research that will guide the evidence-based management of RSE while also providing novel insights into the sensorimotor underpinnings of speech. The central hypothesis is that biofeedback will yield greater gains in speech accuracy than traditional treatment, and that individual deficit profiles will predict relative response to visual-acoustic vs ultrasound biofeedback. This study will enroll n = 118 children who misarticulate the /r/ sound, the most common type of RSE. This first component of the study will evaluate the efficacy of biofeedback relative to traditional treatment in a well-powered randomized controlled trial. Ultrasound and visual-acoustic biofeedback, which have similar evidence bases, will be represented equally.

DETAILED DESCRIPTION:
Randomized Trial Component: Previous findings suggest that biofeedback interventions can outperform traditional speech therapy for children with RSE, but the research base to date is limited to small-scale studies that do not reach the level of evidence needed to support large-scale changes in practice. The primary objective of the C-RESULTS RCT is to test the working hypothesis that a group of individuals randomly assigned to receive biofeedback-enhanced treatment will show larger and/or faster gains in /r/ production accuracy than an equivalent group receiving the same dose of non-biofeedback treatment. To test this hypothesis, n=110 children will be randomly assigned to receive a standard course of intervention with or without biofeedback. Acoustic and perceptual measures will be used to test for differences in both short-term learning of treated targets (Acquisition) and longer-term carryover of learning to untreated contexts (Generalization). In addition, a survey assessing participants' socio-emotional well-being will be collected from caregivers both pre and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 9;0 and 15;11 years of age at the time of enrollment.
* Must speak English as the dominant language (i.e., must have begun learning English by age 2, per parent report).
* Must speak a rhotic dialect of English.
* Must pass a pure-tone hearing screening at 20 decibels Hearing Level (HL).
* Must pass a brief examination of oral structure and function.
* Must exhibit less than thirty percent accuracy, based on trained listener ratings, on a probe list eliciting /r/ in various phonetic contexts at the word level.

Exclusion Criteria:

* Must not receive a T score more than 1.3 standard deviations (SD) below the mean on the Wechsler Abbreviated Scale of Intelligence-2 (WASI-2) Matrix Reasoning.
* Must not receive a standard score below 80 on the Core Language Index of the Clinical Evaluation of Language Fundamentals-5 (CELF-5).
* Must not exhibit voice or fluency disorder of a severity judged likely to interfere with the ability to participate in study activities.
* Must not have an existing diagnosis of developmental disability or major neurobehavioral syndrome such as cerebral palsy, Down Syndrome, or Autism Spectrum Disorder, or major neural disorder (e.g., epilepsy, agenesis of the corpus callosum) or insult (e.g., traumatic brain injury, stroke, or tumor resection).
* Must not show clinically significant signs of apraxia of speech or dysarthria.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Montclair State University, Bloomfield, New Jersey
  - Syracuse University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Preston JL, McCabe P, Tiede M, Whalen DH. Tongue shapes for rhotics in school-age children with and without residual speech errors. Clin Linguist Phon. 2019;33(4):334-348. doi: 10.1080/02699206.2018.1517190. Epub 2018 Sep 10. PMID 30199271
- [Background] Preston JL, McAllister T, Phillips E, Boyce S, Tiede M, Kim JS, Whalen DH. Treatment for Residual Rhotic Errors With High- and Low-Frequency Ultrasound Visual Feedback: A Single-Case Experimental Design. J Speech Lang Hear Res. 2018 Aug 8;61(8):1875-1892. doi: 10.1044/2018_JSLHR-S-17-0441. PMID 30073249
- [Background] Dugan SH, Silbert N, McAllister T, Preston JL, Sotto C, Boyce SE. Modelling category goodness judgments in children with residual sound errors. Clin Linguist Phon. 2019;33(4):295-315. doi: 10.1080/02699206.2018.1477834. Epub 2018 May 24. PMID 29792525
- [Background] Preston JL, Holliman-Lopez G, Leece MC. Do Participants Report Any Undesired Effects in Ultrasound Speech Therapy? Am J Speech Lang Pathol. 2018 May 3;27(2):813-818. doi: 10.1044/2017_AJSLP-17-0121. PMID 29546269
- [Background] Preston JL, McAllister Byun T, Boyce SE, Hamilton S, Tiede M, Phillips E, Rivera-Campos A, Whalen DH. Ultrasound Images of the Tongue: A Tutorial for Assessment and Remediation of Speech Sound Errors. J Vis Exp. 2017 Jan 3;(119):55123. doi: 10.3791/55123. PMID 28117824
- [Background] Preston JL, Leece MC, Maas E. Motor-based treatment with and without ultrasound feedback for residual speech-sound errors. Int J Lang Commun Disord. 2017 Jan;52(1):80-94. doi: 10.1111/1460-6984.12259. Epub 2016 Jun 14. PMID 27296780
- [Background] Campbell H, Harel D, Hitchcock E, McAllister Byun T. Selecting an acoustic correlate for automated measurement of American English rhotic production in children. Int J Speech Lang Pathol. 2018 Nov;20(6):635-643. doi: 10.1080/17549507.2017.1359334. Epub 2017 Aug 10. PMID 28795872
- [Background] Campbell H, McAllister Byun T. Deriving individualised /r/ targets from the acoustics of children's non-rhotic vowels. Clin Linguist Phon. 2018;32(1):70-87. doi: 10.1080/02699206.2017.1330898. Epub 2017 Jul 13. PMID 28703653
- [Background] McAllister Byun T. Efficacy of Visual-Acoustic Biofeedback Intervention for Residual Rhotic Errors: A Single-Subject Randomization Study. J Speech Lang Hear Res. 2017 May 24;60(5):1175-1193. doi: 10.1044/2016_JSLHR-S-16-0038. PMID 28389677
- [Background] McAllister Byun T, Tiede M. Perception-production relations in later development of American English rhotics. PLoS One. 2017 Feb 16;12(2):e0172022. doi: 10.1371/journal.pone.0172022. eCollection 2017. PMID 28207800
- [Background] McAllister Byun T, Campbell H. Differential Effects of Visual-Acoustic Biofeedback Intervention for Residual Speech Errors. Front Hum Neurosci. 2016 Nov 11;10:567. doi: 10.3389/fnhum.2016.00567. eCollection 2016. PMID 27891084
- [Background] McAllister Byun T, Halpin PF, Szeredi D. Online crowdsourcing for efficient rating of speech: a validation study. J Commun Disord. 2015 Jan-Feb;53:70-83. doi: 10.1016/j.jcomdis.2014.11.003. Epub 2014 Dec 15. PMID 25578293
- [Background] Hitchcock ER, Byun TM, Swartz M, Lazarus R. Efficacy of Electropalatography for Treating Misarticulation of /r/. Am J Speech Lang Pathol. 2017 Nov 8;26(4):1141-1158. doi: 10.1044/2017_AJSLP-16-0122. PMID 28834534
- [Background] Harel D, Hitchcock ER, Szeredi D, Ortiz J, McAllister Byun T. Finding the experts in the crowd: Validity and reliability of crowdsourced measures of children's gradient speech contrasts. Clin Linguist Phon. 2017;31(1):104-117. doi: 10.3109/02699206.2016.1174306. Epub 2016 Jun 7. PMID 27267258
- [Background] Hitchcock ER, Harel D, Byun TM. Social, Emotional, and Academic Impact of Residual Speech Errors in School-Aged Children: A Survey Study. Semin Speech Lang. 2015 Nov;36(4):283-94. doi: 10.1055/s-0035-1562911. Epub 2015 Oct 12. PMID 26458203
- [Background] Hitchcock ER, Byun TM. Enhancing generalisation in biofeedback intervention using the challenge point framework: a case study. Clin Linguist Phon. 2015 Jan;29(1):59-75. doi: 10.3109/02699206.2014.956232. Epub 2014 Sep 12. PMID 25216375
- [Background] Byun TM, Hitchcock ER, Swartz MT. Retroflex versus bunched in treatment for rhotic misarticulation: evidence from ultrasound biofeedback intervention. J Speech Lang Hear Res. 2014 Dec;57(6):2116-30. doi: 10.1044/2014_JSLHR-S-14-0034. PMID 25088034
- [Background] Byun TM, Hitchcock ER. Investigating the use of traditional and spectral biofeedback approaches to intervention for /r/ misarticulation. Am J Speech Lang Pathol. 2012 Aug;21(3):207-21. doi: 10.1044/1058-0360(2012/11-0083). Epub 2012 Mar 21. PMID 22442281
- [Derived] McAllister T, Preston JL, Hitchcock ER, Hill J. Protocol for Correcting Residual Errors with Spectral, ULtrasound, Traditional Speech therapy Randomized Controlled Trial (C-RESULTS RCT). BMC Pediatr. 2020 Feb 11;20(1):66. doi: 10.1186/s12887-020-1941-5. PMID 32046671

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Traditional Articulation Treatment: Traditional articulation treatment
- Group 2: Biofeedback--visual-acoustic: Biofeedback--visual-acoustic
- Group 3: Biofeedback-Ultrasound: Biofeedback-ultrasound
Period: Phase 1 (Acquisition)
Arm/Group | Group 1: Traditional Articulation Treatment | Group 2: Biofeedback--visual-acoustic | Group 3: Biofeedback-Ultrasound
Started | 45 | 32 | 31
Primary Outcome Assessment | 45 | 32 | 31
Completed | 45 | 32 | 31
Not Completed | 0 | 0 | 0
Period: Phase 2 (Generalization)
Arm/Group | Group 1: Traditional Articulation Treatment | Group 2: Biofeedback--visual-acoustic | Group 3: Biofeedback-Ultrasound
Started | 45 | 32 | 31
Secondary Outcome Assessment | 45 | 32 | 31
Completed | 41 | 31 | 30
Not Completed | 4 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Traditional Articulation Treatment | Group 2: Biofeedback--visual-acoustic | Group 3: Biofeedback-Ultrasound | Total
Number analyzed (Participants) | 45 | 32 | 31 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.72 (1.54) | 10.86 (1.87) | 10.71 (1.3) | 10.8 (1.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 9 | 40
  Male | 30 | 16 | 22 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 36 | 31 | 27 | 94
  More than one race | 5 | 0 | 1 | 6
  Unknown or Not Reported | 3 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 3 | 8
  Not Hispanic or Latino | 40 | 29 | 25 | 94
  Unknown or Not Reported | 1 | 2 | 3 | 6
Response to dynamic assessment session [Count of Participants; unit: Participants] — Prior to randomization, participants completed a dynamic assessment (DA) session to evaluate their ability to respond to treatment. Participants were categorized into two groups based on the treating clinician's perceptual ratings of their articulation. The two groups were termed high initial responders (greater than 5% accuracy during DA) or low initial responders (0%-5% accuracy during DA). Randomization was stratified by DA response group.
  Participants
    High initial responders | 21 | 14 | 15 | 50
    Low initial responders | 24 | 18 | 16 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in F3-F2 Distance (Hz) Across Sessions, Measured From /r/ Sounds Produced in Syllables or Words During Practice.
Description: F3-F2 distance is a number (in Hz) that reflects how close a child's /r/ sound is to a typical adult-like /r/. Smaller numbers indicate more accurate /r/ production; larger numbers indicate a distorted /r/. In typical peers, accurate /r/ is roughly ~500 Hz, whereas distorted /r/ values are often >1000 Hz. During Phase I (3 sessions over ~1 week), children produced /r/ in syllables/words. For this Outcome, we report change across sessions: a single model-based estimate of how much F3-F2 decreased from Session 1 to Session 3 (i.e., the rate of improvement). A more negative change indicates greater improvement.
Time Frame: Phase I: three 90-min treatment sessions delivered over ~1 week; reported value is the change from Session 1 to Session 3 (slope across sessions)
Population: Three participants from group 2 (visual-acoustic biofeedback) could not be acoustically analyzed due to poor audio quality.
Measure: Mean (Standard Deviation); unit: Hertz / session
Arm/Group | Group 1: Traditional Articulation Treatment | Group 2: Biofeedback--visual-acoustic | Group 3: Biofeedback-Ultrasound
Number analyzed (Participants) | 45 | 29 | 31
Hertz / session | 38.2 (66.0) | 66.7 (103.0) | 85.2 (152.0)
Statistical Analysis 1: Comparison: Group 1: Traditional Articulation Treatment vs Group 2: Biofeedback--visual-acoustic vs Group 3: Biofeedback-Ultrasound; Following our preregistered statistical analysis plan, the visual-acoustic and ultrasound biofeedback groups were pooled for comparison of biofeedback versus traditional treatment; Test type: Superiority; p < .0001, Regression, Linear — Two-sided test of the treatment × time interaction. Alpha = 0.05; Treatment × Time interaction (β) = 106.41, 95% CI 2-sided [63.06 to 149.76], Standard Error of Mean 22.11 — Sign convention: A more positive β indicates a more positive Session 1→3 slope in the traditional treatment group relative to the biofeedback group (reference level)

2. Secondary Outcome: Change From Pre to Post in Percent "Correct" Ratings by Untrained Listeners, for /r/ Sounds Produced in Word Probes.
Description: The outcome is the percentage of untrained listeners, blinded to time point and treatment condition, who judged each /r/ production as "correct" from word-probe recordings (0-100%; higher = better). Children completed word probes at Pre and Post. Results in the table summarize change from Pre to Post using a mixed-effects model: specifically, the treatment × time interaction, which estimates the between-group difference in improvement from Pre to Post. A positive change indicates improvement.
Time Frame: Pre (before initiation of treatment) and Post (after the end of all treatment; ~10 weeks later).
Population: The analysis population differs from the number of participants who completed the Secondary Outcome Assessment visit (Phase 2) because two participants contributed unusable secondary-outcome data (one due to corrupted audio files, and one who completed all treatment sessions but whose number of trials completed did not pass the threshold for inclusion in the analysis).
Measure: Mean (Standard Deviation); unit: Percent words rated correct
Arm/Group | Group 1: Traditional Articulation Treatment | Group 2: Biofeedback--visual-acoustic | Group 3: Biofeedback-Ultrasound
Number analyzed (Participants) | 41 | 30 | 29
Percent words rated correct | 44.5 (34) | 43.2 (33) | 49.6 (34)
Statistical Analysis 1: Comparison: Group 1: Traditional Articulation Treatment vs Group 2: Biofeedback--visual-acoustic vs Group 3: Biofeedback-Ultrasound; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Regression, Linear — Two-sided test of the treatment × time interaction. Alpha = 0.05; Test of treatment × time (Pre, Post) interaction; Treatment × Time (linear) interaction (β = -3.12, 95% CI 2-sided [-4.85 to -1.40], Standard Error of Mean 0.88 — Sign convention: Negative β indicates a smaller linear time slope in the traditional treatment group relative to the biofeedback group (reference level)

3. Secondary Outcome: Impact of Speech Disorder on Social, Emotional, and Academic Well-being (Parent Survey)
Description: Parents completed a questionnaire assessing the impact of their child's speech disorder on social, emotional, and academic well-being. Each item was rated on a 5-point scale (1 = strongly disagree, 3 = neutral, 5 = strongly agree). Scores were averaged across items to yield an overall impact score ranging from 1 to 5, with higher values indicating a greater negative impact. A decrease from Pre to Post indicates improvement.
Time Frame: Pre (before initiation of treatment) and Post (after completion of all treatment; ~10 weeks later)
Population: The number of participants analyzed for secondary outcome measure #3 is the same as the number of participants who completed Phase 2. The data quality-related exclusions that impacted the secondary outcome measure #2 did not impact secondary outcome measure #3.
Measure: Mean (Standard Deviation); unit: Impact score
Arm/Group | Group 1: Traditional Articulation Treatment | Group 2: Biofeedback--visual-acoustic | Group 3: Biofeedback-Ultrasound
Number analyzed (Participants) | 41 | 31 | 30
Impact score | 1.9 (1.1) | 1.9 (1.1) | 2.1 (1.2)
Statistical Analysis 1: Comparison: Group 1: Traditional Articulation Treatment vs Group 2: Biofeedback--visual-acoustic vs Group 3: Biofeedback-Ultrasound; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .80, Regression, Linear — Two-sided test of the treatment × time interaction. Alpha = 0.05; Test of treatment (Traditional vs biofeedback) × linear time; Treatment × Time linear interaction (β) = 0.0147, 95% CI 2-sided [-0.10 to 0.13], Standard Error of Mean 0.0594 — Sign convention: positive β indicates a larger linear time slope in the traditional group relative to the biofeedback group (reference level)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, roughly 13 weeks"
Description: This was a low-risk behavioral speech therapy trial. Adverse events were systematically monitored with safety checks at midpoint and end of treatment. Because all randomized participants were included in adverse event monitoring, all randomized participants were treated as at risk. Study definitions were consistent with ClinicalTrials.gov definitions.
Arm/Group | Group 1: Traditional Articulation Treatment | Group 2: Biofeedback--visual-acoustic | Group 3: Biofeedback-Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/45 | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03737318/Prot_SAP_000.pdf